CLINICAL TRIAL: NCT06325709
Title: Phase 1/2 Trial of Base Editing for Mutation Repair in Hematopoietic Stem & Progenitor Cells for X-linked Chronic Granulomatous Disease
Brief Title: Base Editing for Mutation Repair in Hematopoietic Stem & Progenitor Cells for X-Linked Chronic Granulomatous Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001580; 001580-I
Record Dates: First submitted 2024-03-21; First posted 2024-03-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Chronic Granulomatous Disease (CGD); X-Linked Chronic Granulomatous Disease
Keywords: base editing; Gene Editing
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — plerixafor; Filgrastim; Fibroblast Growth Factor 7; Busulfan; Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental)
  Interventions: Drug: Plerixafor; Drug: Filgrastim; Drug: Palifermin; Drug: Busulfan; Biological: Base-edited hematopoietic stem and progenitor cells; Drug: Sirolimus

INTERVENTIONS:
Drug: Plerixafor — Stem Cell Mobilizing Agent: Subcutaneous administration for 2 consecutive days to improve stem cell collection.
Drug: Filgrastim — Stem Cell Mobilizing Agent: Subcutaneous administration for 6 consecutive days. It is necessary to mobilize stem cells for collection.
Drug: Palifermin — Mucositis Prophylaxis Agent: Intravenous infusion of keratinocyte growth factor (Palifermin) at 60 mcg/kg/day before (Days -7 to Day -5 administration of busulfan and (Days 1 to 3) post-busulfan administration to prevent oral mucositis.
Drug: Busulfan — Transplant Conditioning Agent: An alkylating chemotherapy drug to enhance engraftment of the study agent (base-edited stem cells). Conditioning will be given intravenously over 3 days with an approximate total dose of 12mg/kg. Drug levels obtained will be obtained to achieve the targeted total busulfan AUC of 65,000 ng/mL x hr.
Biological: Base-edited hematopoietic stem and progenitor cells — Investigational/Study Agent: Base-edited autologous CD34 plus hematopoietic stem and progenitor cell product. The product is administered intravenously as a single infusion. This product is under an IND.
Drug: Sirolimus — Immunomodulating agent: Daily oral dosing beginning Day -1 for approximately 3 to 6 months to prevent an immune response to the protein expressed by the BE HSPCs.

SUMMARY:
Background:

Chronic granulomatous disease (CGD) is a rare immune disorder caused by a mutation in the CYBB gene. People with CGD have white blood cells that do not work properly and are at greater risk of getting infections. Gene therapy using lentivector has helped people with CGD. Researchers want to know if the base-edited stem cells can improve the white cells' functioning and result in fewer CGD-related infections.

Objective:

To learn if base-edited stem cells will correct the white blood cells in people with CGD.

Eligibility:

Males aged 18 years and older with X-linked CGD.

Design:

This is a non-randomized study. Participants with the specific mutation under study will be screened during the initial phase.

During the development phase, participants will undergo apheresis to collect stem cells for base-editing correction of the mutation.

During the treatment phase, participants will receive the base-edited cells after chemotherapy with busulfan. Participants will remain in the hospital until their immunity recovers. Participants will be maintained on sirolimus to prevent an immune response to the new protein expressed by the base-edited cells.

Follow-up visits will continue for 15 years....

DETAILED DESCRIPTION:
Study Description:

Open-label, phase 1/2 trial to determine the safety, and efficacy of a single infusion of base-edited (BE) autologous hematopoietic stem and progenitor cells (HSPCs) for treatment of X-linked chronic granulomatous disease (X-CGD). Base editing is performed to repair CYBB missense gene mutations (eg, CYBB c.676C>T). The study hypotheses are that 1) base editing can efficiently repair gene mutations in HSPCs; and 2) BE HSPCs can engraft and differentiate into functional phagocytes with restored nicotinamide adenine dinucleotide phosphate (NADPH) oxidase activity.

During the initial development phase each study participant will undergo apheresis for CD34+ HSPC collection for the development and validation of a mutation-specific BE system.

During the treatment phase, participants will receive a one-time infusion of the BE autologous HSPC (study product) after the administration of busulfan conditioning (total 12 mg/kg with a targeted total AUC of 65,000 ng/mL x hr). Sirolimus will be initiated at Day -1 and will be given for approximately 3-6 months.

Participants will have follow-up evaluations at months 3, 6, 12, 18, and 24, and yearly thereafter until 5 years after treatment. Key study assessments include adverse event (AE) assessment, blood laboratory evaluations of functional protein made from the target gene (CYBB, encodes for gp91^phox), and deoxyribonucleic acid (DNA) sequencing to identify rates of gene repair and off-target mutation.

The final study follow-up under this protocol will be at 5 years, but long-term follow-up under a separate NIH protocol will continue annually to 15 years after treatment.

Objectives:

Primary Objectives:

* To evaluate the safety of BE autologous CD34+ cells.
* To evaluate the efficacy of BE autologous CD34+ cells.

Secondary Objectives:

-To evaluate:

* Efficiency of base editing (percentages of target nucleotide conversion).
* Engraftment capability of BE HSPCs.
* Efficiency in restoring gp91^phox expression
* Efficiency in restoring NADPH oxidase function.
* Clinical efficacy.
* Stability of gene correction.

Exploratory Objectives:

-To evaluate:

* Specificity of base editing by assessing rates of off-target edits at top predicted sites.
* Random off-target edits by whole genome sequencing (WGS).

Endpoints:

Primary Endpoints:

* Safety of gene therapy using BE autologous HSPCs as measured by study product-related AEs and serious AEs (SAEs) through 2 years after treatment.
* Efficacy of gene therapy determined as percentages of subjects who have >= 10% oxidase-positive granulocytes at 12 months after infusion.

Secondary Endpoints:

* Determine frequency of converted target nucleotide alleles.
* Assess the frequency of gene-modified alleles compared to infusion product in peripheral blood at 12 months.
* Evaluate efficacy of restoring gp91^phox expression.
* Evaluate efficacy of NADPH oxidase functional restoration as measured by the dihydrorhodamine (DHR) flow cytometry oxidase assay at 12 months after treatment (>=10% oxidase-positive neutrophils), or by quantitative measurement of reactive oxygen species (ROS) using the ferricytochrome C assay on peripheral blood granulocytes.
* Evaluate clinical benefit by improvement of baseline clinical problems such as recurrent infections, growth failure, malnutrition, inflammatory bowel disease, or antibiotic usage.
* Assess stability of gene correction by serial measurement of percent of nucleotide-converted alleles.

Exploratory Endpoints:

* Evaluate specificity by assessing for off-target edits at predicted sites with high-throughput sequencing of the 5 most common candidate off-target loci identified by a comprehensive in vitro screen, Circularization for High-throughput Analysis of Nuclease Genome-wide Effects by sequencing (CHANGE-seq-BE), in peripheral blood cells.
* Determine rate of random off-target edits WGS.

ELIGIBILITY:
* INCLUSION CRITERIA:

  ->= 18 years of age.
* Confirmed CYBB c.676 C>T mutation.
* Male patients.
* Clinically stable and eligible to undergo apheresis and conditioning chemotherapy.

  ->=5 x 10^6 cryopreserved cells/kg body weight available for study product manufacturing.
* History of at least one prior serious infection or inflammatory complication requiring hospitalization despite conventional therapy.
* In the experience of a qualified clinical investigator, the patient has a poor prognosis.
* Able and willing to use a highly effective method of contraception, AND partner has communicated her willingness through subject to do same, if engaging in potentially reproductive sex from the signing of the informed consent and for 6 months after IMP infusion. Acceptable methods of contraception include the following:

  * Hormonal contraception in continuously effective use by female partner.
  * Male or female condom with spermicide as indicated.
  * Diaphragm or cervical cap in consistent and effective pattern of use with a spermicide by female partner.
  * Intrauterine device in-situ throughout above period by female partner.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

* Untreated, acute infection.
* Elevated anti-gp91 specific autoantibodies >2 x ULN
* Elevated anti-gp91 specific T cells (>10 fold)
* Anti-platelet antibody screening with >1 anti-platelet antibody positive in the presence of an ongoing brain infection; OR >1 anti-platelet antibody positive and considered unsafe for study participation after consultation with hematology specialist.
* Known hypersensitivity to busulfan or any component of the product.
* Contraindications for administration of busulfan.
* Any current or pre-existing hematologic malignancy.
* Chronic infections that are considered unsafe for participation in the study by Infectious Disease Consultant.
* Cardiac abnormalities and neurological abnormalities that are deemed unsafe to participate in the study.
* Childhood malignancy (occurring before 18 years of age) in the patient or a first degree relative, or previously diagnosed known genotype of the participant conferring a predisposition to cancer (no DNA or other testing for cancer predisposition genes will be performed as part of the screen for this protocol).
* Hematological parameters unsafe for apheresis or above Grade 2 Common Terminology Criteria for Adverse Events (CTCAE) criteria until improved.
* Hepatic dysfunction- alanine aminotransferase (ALT >3.0 - 5.0 x upper limit of normal [ULN]), aspartate aminotransferase (AST >3.0 - 5.0 x ULN), bilirubin (>1.5 - 3.0 x ULN).
* Renal dysfunction-serum creatinine >1.5 - 3.0 x ULN or creatinine clearance 59-30 mL/min/1.73 m^2.
* Coagulation dysfunction- Prothrombin INR or Partial thromboplastin time >2 x ULN (patients on controlled anticoagulation agents will not be excluded for therapeutic levels).
* Uncontrolled hypertension- Systolic BP 140-159 mm Hg or diastolic BP 90-99 mm Hg.
* Abnormal blood chemistries- Hyperkalemia (K >5.5 - 6.0 mmol/L), Hypokalemia (<LLN - 3.0 mmol/L and requiring intervention); OR Hypercalcemia (corrected serum calcium >11.5 - 12.5 mg/dL), Hypocalcemia (corrected serum calcium <8.0 -7.0 mg/dL)

These values exclude false abnormalities secondary to hemolysis.

* Cytogenetic abnormalities evidenced on bone marrow aspirate.
* Pulmonary dysfunction FEV1<25% predicted.
* Previous treatment with gene therapy or gene editing products.
* Previous receipt of non-HLA matched donor granulocyte transfusions.
* Any other condition that, in the opinion of the investigator, may unduly compromise the safety or compliance of the patient, or would make successful study completion highly unlikely.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of base-edited autologous CD34+ cells | Initiated from the time of the infusion of base-edited cells through 2 years post-infusion
  Safety of gene therapy using base-edited autologous hematopoietic stem and progenitor cells as measured by study agent related adverse events and serious adverse events
To evaluate the efficacy of base-edited autologous CD34+ cells | Assessed 12 months post-infusion of base-edited cells
  Efficacy of gene therapy as determined by percentages ofparticipants who have >= 10 percent oxidase-positive granulocytes

SECONDARY OUTCOMES:
Evaluate the efficiency of base-editing. | Assessed 12-24 months post-infusion of base-edited cells
  Measure the percentages of gp91-expressing cells
Evaluate the engraftment capability of base-edited hematopoietic stem progenitor cells. | Assessed 12-24 months post-infusion of base-edited cells
  Measure the percentages of edited myeloid cells
Evaluate the efficiency in restoring gp91phox expression. | Assessed 12-24 months post-infusion of base-edited cells
  Measure the frequency of gp91phox+ cells and the amount of gp91phox protein
Evaluate efficacy in restoring NADPH oxidase function. | Assessed 12-24 months post-infusion of base-edited cells
  Measure the frequency of DHR+ cells
Evaluate clinical efficacy | Assessed through study completion
  Assess the frequency of infections and progression of co-morbidities of CGD
Evaluate the stability of gene correction | Assessed through study completion
  Compare frequencies of corrected alleles before infusion and at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Suk S De Ravin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Komor AC, Badran AH, Liu DR. Editing the Genome Without Double-Stranded DNA Breaks. ACS Chem Biol. 2018 Feb 16;13(2):383-388. doi: 10.1021/acschembio.7b00710. Epub 2017 Oct 9. PMID 28957631
- [Background] Kuhns DB, Alvord WG, Heller T, Feld JJ, Pike KM, Marciano BE, Uzel G, DeRavin SS, Priel DA, Soule BP, Zarember KA, Malech HL, Holland SM, Gallin JI. Residual NADPH oxidase and survival in chronic granulomatous disease. N Engl J Med. 2010 Dec 30;363(27):2600-10. doi: 10.1056/NEJMoa1007097. PMID 21190454
- [Derived] Bzhilyanskaya V, Ma L, Liu S, Fox LR, Whittaker MN, Meis RJ, Choi U, Lawson A, Ma M, Theobald N, Burkett S, Sweeney CL, Lazzarotto CR, Tsai SQ, Lack JB, Wu X, Dahl GA, Malech HL, Kleinstiver BP, De Ravin SS. High-fidelity PAMless base editing of hematopoietic stem cells to treat chronic granulomatous disease. Sci Transl Med. 2024 Oct 16;16(769):eadj6779. doi: 10.1126/scitranslmed.adj6779. Epub 2024 Oct 16. PMID 39413163
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001580-I.html